CLINICAL TRIAL: NCT06428682
Title: Role of Intravenous Tranexamic Acid Use in Patients Undergoing Breast Free Flap Reconstruction: Randomized Controlled Trial
Brief Title: Role of TXA in Patients Undergoing Breast Free Flap Reconstruction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John Stranix, Assistant Professor of Plastics Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR220370
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Blood Loss, Surgical
Keywords: Autologous breast reconstruction; Free Flap; Tranexamic Acid
MeSH Terms: conditions — Breast Neoplasms; Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TXA group (Experimental): Women undergoing immediate or delayed free flap breast reconstruction and receiving IV TXA
  Interventions: Drug: Tranexamic acid
- Placebo group (Placebo Comparator): Women undergoing immediate or delayed free flap breast reconstruction and receiving same volume of IV saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Experimental group will receive TXA intraoperatively (15mg/kg IV, once at beginning of case then re dose at 4hrs if operation goes longer) at the time of their surgery.
  Arms: TXA group
Drug: Placebo — Control group will receive same volume equivalent of saline intravenously at the time of their surgery.
  Arms: Placebo group

SUMMARY:
Tranexamic acid (TXA) is a synthetic, competitive lysine receptor inhibitor on plasminogen. It ultimately stabilizes the fibrin matrix, therefore used as a hemostatic agent for various indications. While there has been indications for orthopedic and trauma surgery, there is no clear data for its role in patients who are undergoing free tissue transfer. Studies have shown that patients undergoing free tissue transfer can have transfusion rates ranging from 7.2% to 34.9%, which data also showing association between transfusion requirement and higher free flap failure rate. There has been a few retrospective studies that evaluated the effect of TXA in free tissue transfer and the results showed no increased risk of microanastomosis failure but some showing decreased blood loss. This study aims to further analyze the role of TXA in patients undergoing breast free flap reconstruction with randomized, prospective trial. Control group will not receive TXA while experimental group will receive TXA. Both groups will receive standard of care breast free flap surgery as well as post-op care, which is streamlined with Early Recovery After Surgery (ERAS) protocol. Their pre and post-op hemoglobin will be compared, as well as rates of transfusion, surgical outcome and surgical complications including hematoma, flap failure, and any other medical complications such as Deep Vein Thrombosis (DVT)/ Pulmonary Embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* All female patients who are 18 years or older who will undergo unilateral or bilateral abdomen-based free flap breast reconstruction at UVA Medical Center

Exclusion Criteria:

* Subjects with ages <18 years
* Allergy to TXA
* Subjects who has contraindications to TXA: anyone who has active intravascular thrombosis or anyone with subarachnoid hemorrhage
* Subjects who have anemia (defined as baseline hemoglobin <8 g/dL
* Subjects who cannot read or understand English
* Subjects who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Delta Hemoglobin | 1 day after surgery
  Post-op day 1 Hemoglobin - Pre-op Hemoglobin
Transfusion rate | Typically 0-72 hours after surgery
  Transfusion rate during hospital stay

SECONDARY OUTCOMES:
Surgical complications | 30 days after surgery
  Thromboembolic event, hematoma, seroma, flap compromise/ failure
Length of Stay | typically 2-4 days
  Total length of stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Stranix, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States